CLINICAL TRIAL: NCT00039351
Title: Diffuse Large B Cell And Peripheral T-Cell Non-Hodgkin's Lymphoma In The Frail Elderly. Progressive And Cautious Treatment Strategy In Poor Status Patients. A Phase II Trial With Emphasis On Geriatric Assessment And Quality Of Life
Brief Title: Combination Chemotherapy in Treating Older Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-20992; EORTC-20992
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; angioimmunoblastic T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Immunoblastic Lymphadenopathy | interventions — Cyclophosphamide; Prednisone; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating older patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete remission (CR) rate and duration of CR in frail elderly patients with diffuse large B-cell or peripheral T-cell non-Hodgkin's lymphoma treated with cyclophosphamide, vincristine, and prednisone.
* Determine the time to progression and overall survival of patients treated with this regimen.
* Determine the severe toxicity rate of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive cyclophosphamide IV and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients with stage I or II non-Hodgkin's lymphoma (NHL), no baseline lactate dehydrogenase (LDH) elevation, baseline WHO performance status 0-1, and longest tumor diameter of less than 5 cm, who achieve partial response (PR) or complete response (CR), receive 1 additional course of chemotherapy. Patients then undergo involved-field radiotherapy once daily 5 days a week for 3.5-4 weeks.

Patients with stage I or II NHL, a baseline LDH elevation, and/or baseline WHO performance status 2-4, and/or longest tumor diameter of at least 5 cm, who achieve PR or CR, receive 3 additional courses of chemotherapy. Patients then undergo involved-field radiotherapy once daily 5 days a week for 3.5-4 weeks.

Patients with stage III or IV NHL who achieve CR or PR receive 3 additional courses of chemotherapy. Patients then undergo consolidative radiotherapy once daily 5 days a week for 2.5-3 weeks.

Quality of life is assessed at baseline, after the third chemotherapy course, at the end of chemotherapy, every 6 months for 3 years, and then annually thereafter.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 29-56 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large B-cell or peripheral T-cell non-Hodgkin's lymphoma (NHL)

  * No Burkitt's-like lymphoma
  * Small cells in bone marrow allowed
* Previously untreated NHL
* At least 1 measurable lesion

  * At least 1.1 cm
* Poor physiological status with at least 1 of the following:

  * WHO performance status of 3-4
  * LVEF less than 50%
  * Creatinine clearance less than 50 mL/min
  * Neutrophil count no greater than 1,500/mm^3
  * Platelet count no greater than 100,000/mm^3
  * Concurrent severe disease that would preclude cyclophosphamide, vincristine, prednisolone, and doxorubicin
* No cerebral or meningeal involvement

PATIENT CHARACTERISTICS:

Age:

* 70 and over

Performance status:

* See Disease Characteristics

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* See Disease Characteristics

Other:

* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell skin cancer, curatively treated carcinoma in situ of the cervix, or curatively treated solid tumor
* No active infection
* No psychological, familial, sociological, or geographical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent investigational drugs
* No other concurrent antineoplastic agents

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-03; Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Soubeyran, MD, PhD, Study Chair — Institut Bergonié
Locations (17):
- Belgium (3):
  - Ziekenhuis Network Antwerpen Middelheim, Antwerp
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - U.Z. Gasthuisberg, Leuven
- National Cancer Institute of Egypt, Cairo, Egypt
- France (6):
  - Centre D'Oncologie Du Pays-Basque, Bayonne
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier de Dax, Dax
  - Hopital Robert Boulin, Libourne
  - Polyclinique de Francheville, Périgueux
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Hopitaux Universitaires de Geneve, Thonex-Geneve, Switzerland
- United Kingdom (2):
  - New Cross Hospital, Wolverhampton, England
  - Dumfries Royal Infirmary, Dumfries